CLINICAL TRIAL: NCT02033174
Title: Effects of Acute and Chronic Red Wine Intake in the Expression of Pro-inflammatory and Prothrombotic Factors in Circulating Monocytes
Brief Title: Effects of Alcoholic Beverages in Pro-inflammatory and Antioxidant Profile After an Oral Fat Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Gregorio Marañón (Other)
Responsible Party: Principal Investigator, Luis A. Alvarez-Sala, MD, Instituto de Investigación Sanitaria Gregorio Marañón
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AlcoholInfl_IiSGM_2000; FIS01/0602 (Other Grant/Funding Number: Fondo de Investigaciones Sanitarias FIS01/0602.)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Alcohol Consumption
Keywords: alcohol, inflammation, oxidation.
MeSH Terms: conditions — Alcohol Drinking; Inflammation | interventions — Water; Sugars; Alcoholic Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar water first, then alcohol (Other): 8 participants have received oral fat diet plus water with sugar (equivalent caloric intakes as sugar with water in the control group). Then they receive the same oral fat-enriched diet (1486 kcal/m2) with 654 kcal/m2 (44%) as fat and a daily total amount of 16 g/m2 of alcohol, of different beverages (red wine, vodka, brandy or rum)
  Interventions: Other: Oral fat diet plus water with sugar; Other: Oral fat diet plus alcoholic beverages
- Alcohol first then sugar water (Other): 8 participants have received oral fat diet plus alcoholic beverages (a daily total amount of 16 g/m2 of alcohol, of different beverages : red wine, vodka, brandy or rum). Then they receive the same oral fat-enriched diet (1486 kcal/m2) with 654 kcal/m2 (44%) as fat and water with sugar (equivalent caloric intakes as sugar with water in the control group).
  Interventions: Other: Oral fat diet plus water with sugar; Other: Oral fat diet plus alcoholic beverages

INTERVENTIONS:
Other: Oral fat diet plus water with sugar — All participants were assigned to receive and oral fat diet plus sugar water. Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat. Sugar water has equivalent caloric intakes as alcoholic beverages.
Other: Oral fat diet plus alcoholic beverages — Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat. In all cases, alcohol represented a daily total amount of 16 g/m2. The content of alcohol was 12% in red wine, 37% in rum, and 35% in brandy.Vodka was tri-distilled and contained 40% alcohol.

SUMMARY:
Hypothesis: Red wine intake but not other alcoholic beverages together with a fat diet will decrease inflammatory factors and lipid peroxidation and decrease antioxidant capacity in healthy people after a five days period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Individuals with a plasma cholesterol level > 220 mg/dl
* Smokers

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-01; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Alvarez-Sala, PhD, MD, Principal Investigator — Head of section. Dep. of Internal Medicine
Locations (1):
- IiSGM, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol First, Then Sugar Water: Participants first received an oral fat-enriched diet (1486 kcal/m2) and a daily total amount of 16 g/m2 of alcohol, of different beverages (red wine, vodka, brandy or rum) for 5 days. Then, they received equivalent caloric intakes as sugar with water in the control group for 5 days.
- Sugar Water First ,Then Alcohol: Participants first received an oral fat-enriched diet (1486 kcal/m2) and sugar with water for 5 days. They then received a daily total amount of 16 g/m2 of alcohol, of different beverages (red wine, vodka, brandy or rum) for 5 days.
Period: First Intervention
Arm/Group | Alcohol First, Then Sugar Water | Sugar Water First ,Then Alcohol
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Alcohol First, Then Sugar Water | Sugar Water First ,Then Alcohol
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Alcohol First, Then Sugar Water | Sugar Water First ,Then Alcohol
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Cross over study over five different weeks. Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat. In all cases, alcohol represented a daily total amount of 16 g/m2. The content of alcohol was 12% in red wine, 37% in rum, and 35% in brandy.Vodka was tri-distilled and contained 40% alcohol.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Concentrations of Antioxidant Profile After Red Wine Intake
Description: In order to determine total antioxidant capacity a quantitative immunoassay using commercial kits (R&D Systems, Inc. Minneapolis, USA) was conducted.
Time Frame: Baseline and 5 days
Population: All participants who completed all study visits were included
Measure: Median (Inter-Quartile Range); unit: percentage of change in TAC
Groups:
- Alcoholic Beverages (Red Wine Intake): Cross over study over five different weeks. Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat. In all cases, alcohol represented a daily total amount of 16 g/m2. The content of alcohol was 12% in red wine
- Oral Fat Diet: The fat-enriched diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat.
Arm/Group | Alcoholic Beverages (Red Wine Intake) | Oral Fat Diet
Number analyzed (Participants) | 16 | 16
percentage of change in TAC | 22.3 [19.7 to 25.9] | 12.7 [8.1 to 20.3]
Statistical Analysis 1: Comparison: Alcoholic Beverages (Red Wine Intake) vs Oral Fat Diet; Test type: Superiority or Other; p = 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Groups:
- Alcoholic Beverages: Cross over study over five different weeks. Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat. In all cases, alcohol represented a daily total amount of 16 g/m2. The content of alcohol was 12% in red wine, 37% in rum, and 35% in brandy.Vodka was tri-distilled and contained 40% alcohol.
- Oral Fat Diet: Oral fat diet contained 1487 kcal/m2 with 654 kcal/m2 (44%) as fat.
Arm/Group | Alcoholic Beverages | Oral Fat Diet
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No